CLINICAL TRIAL: NCT02464202
Title: Use of Stereolithographic Model in Tooth Autotransplantation and Periodontal Ligament Stem Cells for Pulp Revascularization and Reinnervation to Increase the Success Rate for Tooth Replacement in Children
Brief Title: Use of CBCT-based Tooth Replica in Tooth Autotransplantation to Improve the Outcome of Tooth Replacement in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Research Foundation Flanders (Other)
Responsible Party: Principal Investigator, Reinhilde Jacobs, Prof. Dr., Universitaire Ziekenhuizen KU Leuven
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G089213N
Record Dates: First submitted 2014-12-02; First posted 2015-06-08 (Estimated); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: Increase Success Rate of Tooth Transplantation
Keywords: Tooth autotransplantation; stereolithography tooth replica; CBCT; Outcome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- stereolithography tooth replica (Experimental): stereolithographic tooth replica used as a guide for tooth autotransplantation decreases extra-alveolar time and reduces trauma to periodontal ligament tissue therefore increasing the success rate after transplantation
  Interventions: Other: stereolithography tooth replica

INTERVENTIONS:
Other: stereolithography tooth replica — Tooth replica will be made and used for preparing the receiving tooth socket during autotransplantation

SUMMARY:
The aim of this study lies in comparing the outcome of the proposed technique in a large sample size group to the outcome of the conventional tooth autotransplantation method and to provide sufficient evidence for improving the long-term success rate of the tooth autotransplantation procedure.

ELIGIBILITY:
Inclusion Criteria:

The subjects will be divided in two groups according to different surgical protocols.

1. Pediatric subjects (age between 9-18 years) treated with the CBCT-based replica procedure (prospective approach).

   Pediatric subjects (N=50) that missed their teeth due to agenesis or lost their permanent teeth due to trauma, caries, and endodontic failure and referred to dentistry department for replacement of the missing tooth by means of tooth autotransplantation.
2. Pediatric subjects (age between 9-18 years) treated with the conventional method (prospective and retrospective).

Pediatric subjects (N=50) that missed their teeth due to agenesis or lost their permanent teeth due to trauma, caries, and endodontic failure and referred to dentistry department for replacement of the missing tooth by means of tooth autotransplantation.

A matched control patient will be selected with the focus on a very similar surgical challenge, based on age, gender and a matching donor tooth with the same stage of root development and host bed.

Exclusion Criteria:

* Potential participants (case and control) will be excluded if follow-up data are missing for the one-year follow-up.

Ages: 9 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2013-05; Primary Completion 2016-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
success rate | 5 years
survival rate | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- KULeuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No
Patient is already informed and in follow-up after the surgery.

REFERENCES:
- [Derived] EzEldeen M, Wyatt J, Al-Rimawi A, Coucke W, Shaheen E, Lambrichts I, Willems G, Politis C, Jacobs R. Use of CBCT Guidance for Tooth Autotransplantation in Children. J Dent Res. 2019 Apr;98(4):406-413. doi: 10.1177/0022034519828701. Epub 2019 Feb 20. PMID 30786806